CLINICAL TRIAL: NCT02079168
Title: A Multi-Center, Prospective, Randomized, Single-Blind, Within-Subject Controlled, Phase 2a Study to Evaluate the Effectiveness and Safety of RXI-109 on the Outcome of Keloid Excision Surgery in Healthy Adults
Brief Title: A Study to Evaluate the Effectiveness and Safety of RXI-109 on the Outcome of Keloid Excision Surgery in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RXi Pharmaceuticals, Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RXI-109-1401
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Keloid
Keywords: Keloid; Cicatrix; Keloid prevention; Keloid revision/excision; Keloidectomy
MeSH Terms: conditions — Keloid; Cicatrix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Treatment with RXI-109 at the site of one excised keloid and a placebo at the site of a second excised keloid. Dosing to begin at the time of surgery.
  Interventions: Drug: RXI-109; Drug: Placebo
- Cohort 2 (Experimental): Treatment with RXI-109 at the site of one excised keloid and a placebo at the site of a second excised keloid. Dosing to begin two weeks after surgery.
  Interventions: Drug: RXI-109; Drug: Placebo

INTERVENTIONS:
Drug: RXI-109
Drug: Placebo

SUMMARY:
To evaluate the effectiveness of RXI-109 in reducing the recurrence of keloid formation following elective keloid excision.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 21-55 years of age.
* Two keloids of approximately similar size and anatomical location on the earlobe, neck, or torso.
* Keloids to be excised must have been present for > 1 year.

Exclusion Criteria:

* Use of tobacco or nicotine-containing products
* Pregnant or lactating
* Post-menopausal or full hysterectomy

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Reduction in the recurrence of a keloid after keloid excision | 6 months
  To evaluate the effectiveness of RXI-109 in reducing the recurrence of keloid formation following elective keloid excision

SECONDARY OUTCOMES:
Safety of RXI-109 | 6 months
  To assess severity and frequency of reported adverse events and clinically-relevant changes in laboratory testing after elective excision of a keloid

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Pavco, PhD, Study Director — RXi Pharmaceuticals
Locations (3):
- United States (2):
  - Miami, Florida
  - St Louis, Missouri
- San Cristóbal, Dominican Republic